CLINICAL TRIAL: NCT01941446
Title: A Randomized, Placebo- and Positive Controlled, Three-Way, Crossover Study to Evaluate the Effects of an Intravenous Infusion of Eravacycline (TP-434) on Cardiac Repolarization in Healthy Male and Female Subjects: A Thorough QT/QTc Study
Brief Title: A Thorough QT/QTc Study to Evaluate the Effects of an Intravenous Infusion of Eravacycline (TP-434) on Cardiac Repolarization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP-434-004
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Normal Healthy Subjects
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- pre-generated treatment scheme (Experimental): Treatment A: Eravacycline (TP-434) 1.5 mg/kg administered intravenously over 60 minutes and one placebo oral tablet
  Interventions: Drug: Eravacyline, Moxifloxacin, and placebo
- Pre-generated tratment scheme (Placebo Comparator): Treatment B: Placebo (0.9% sodium chloride) administered intravenously over 60 minutes and one moxifloxacin 400 mg oral tablet
  Interventions: Drug: Eravacyline, Moxifloxacin, and placebo
- Moxifloxacin (Placebo Comparator): Treatment C: Placebo (0.9% sodium chloride) administered intravenously over 60 minutes and one placebo oral tablet
  Interventions: Drug: Eravacyline, Moxifloxacin, and placebo

INTERVENTIONS:
Drug: Eravacyline, Moxifloxacin, and placebo

SUMMARY:
This is a randomized, placebo- and positive-controlled (moxifloxacin), 3-period, 3-way crossover thorough QT study, which includes a Screening Period, Treatment Periods (1 through 3), and a Follow-up Visit. Subjects will be confined to the investigational site for 4 nights/3 days during Period 1 and for 3 nights/2 days during Periods 2 and 3. There will be a minimum of a 14 day washout between treatments.

DETAILED DESCRIPTION:
Each of the following treatments will be evaluated on Day 1 of each period in a crossover fashion. The IV eravacycline (TP-434) and IV placebo will be double-blinded.

* Treatment A: Eravacycline (TP-434) 1.5 mg/kg administered intravenously over 60 minutes and one placebo oral tablet;
* Treatment B: Placebo (0.9% sodium chloride) administered intravenously over 60 minutes and one moxifloxacin 400 mg oral tablet; and
* Treatment C: Placebo (0.9% sodium chloride) administered intravenously over 60 minutes and one placebo oral tablet.

Subjects will be randomized to a treatment sequence according to a pre-generated treatment scheme. Subjects will receive a different treatment during each of the 3 periods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects of 18 to 55 years of age;
2. Females must be surgically sterile (hysterectomy and/or bilateral oophorectomy), post-menopausal for 1 year (with follicle-stimulating hormone [FSH] in menopausal range), or agree to use 2 medically accepted, effective methods of birth control (e.g., hormonal contraception, including oral, implant/patch, or injection, or latex condom with spermicide, diaphragm with intravaginal spermicide, cervical cap with spermicide, or indwelling intrauterine device) from the time of signing informed consent until 2 weeks after the Follow-Up Visit. One of the birth control methods must be a barrier method;
3. Male subjects with sexual partners of childbearing potential must agree to use 2 medically accepted, effective methods of birth control (e.g., hormonal contraception, including oral, implant/patch, or injection, or latex condom with spermicide, diaphragm with intravaginal spermicide, cervical cap with spermicide, or indwelling intrauterine device) for the duration of the study and for 90 days after the Follow-up Visit. Male subjects who have had a vasectomy >6 months prior to the first dose of study drug must agree to use 1 medically accepted barrier method for the duration of the study and for 90 days after the Follow-up Visit;
4. Male subjects (including those who have had vasectomies >6 months prior to the first dose of study drug) whose partners are currently pregnant must agree to use a barrier method (without spermicide) for the duration of the study and for 2 weeks after the Follow-up Visit;
5. Body mass index of 18 kg/m2 to 33 kg/m2, inclusive;
6. Non-smokers must have quit smoking >3 months prior to the Screening Visit;
7. Have negative alcohol and drug screens;
8. Have a quantitative urine cotinine screen <3;
9. Willing and able to be confined to the investigational site as required by the protocol; and
10. Able to comprehend and willing to provide written informed consent in accordance with institutional and regulatory guidelines.

Exclusion Criteria:

1. Evidence of clinically significant hematologic, renal, endocrine, pulmonary, cardiac, gastrointestinal, hepatic, psychiatric, neurologic, or allergic disease (including multiple or clinically significant drug allergies), cancer, or any other condition that, in the opinion of the Investigator, might significantly interfere with the absorption, distribution, metabolism, or excretion of study drug, interfere with the integrity of electrophysiologic data, or place the subject at an unacceptable risk as a participant in this study;
2. A personal or family history of long QT syndrome, Torsades de pointes, or other complex ventricular arrhythmias or family history of sudden death;
3. Mean QTcF interval >450 msec on screening ECG, performed in triplicate. The mean QTcF of these tracings will be used by the Investigator;
4. Cardiac conduction abnormalities denoted by any of the following at the Screening Visit: evidence of second-degree (Mobitz type II) or third-degree atrioventricular block, evidence of ventricular pre-excitation, complete left bundle branch block, right bundle branch block, intraventricular conduction delay with QRS duration >120 msec, atrial fibrillation, or presence of cardiac pacemaker; PR interval >220 msec or <120 msec; heart rate <45 bpm or >90 bpm; other clinically-significant ECG abnormalities (measured as a mean value from triplicate ECGs);
5. Use of hormone replacement therapy;
6. Any major surgical procedure within 3 months prior to the first dose of study drug;
7. Gastrointestinal disorders or surgical procedures that could interfere significantly with the absorption of orally administered drugs;
8. Use of another investigational drug or device within 30 days prior to receiving eravacycline (TP-434), or within at least 5 half-lives of the previous investigational drug, whichever is longer;
9. History of malignancy (other than basal cell or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer);
10. History or presence of hypertension (defined as systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg). If the subject's blood pressure is outside of the acceptable range at the Screening Visit, the subject may be retested within 24 hours at the discretion of the Investigator;
11. Known allergies to moxifloxacin, other quinolone or tetracycline antibiotics, or related compounds or a history of multiple adverse drug allergies of any origin;
12. Inadequate venous access;
13. Obvious clinical signs or symptoms of liver disease, acute or chronic active hepatitis, or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 the upper limit of normal (ULN). An abnormal ALT or AST test may not be repeated;
14. Total bilirubin >1.5 ULN with elevated direct bilirubin. An abnormal total or direct bilirubin test may not be repeated;
15. Serum potassium, magnesium, or calcium levels that are outside of the laboratory's reference range;
16. History of alcoholism or drug abuse within 2 years prior to dosing;
17. Typical weekly alcohol consumption of 14 alcoholic drinks. One drink is defined as 1 glass of beer (approximately 10 oz to 12 oz) or 1 can (12 oz) of beer, 1 glass of wine (approximately 4 oz to 5 oz), or 1 glass of distilled spirits (hard liquor) containing 1 oz of the liquor (1 oz of liquid is approximately 30 mL);
18. Alcohol consumption within 48 hours prior to dosing;
19. Use of tobacco, nicotine, or nicotine-replacement products within the 3 months prior to the first dose of study drug through the last study visit;
20. Unwillingness to refrain from caffeine and other xanthine-containing beverages, including coffee and tea, as well as grapefruit juice, Seville oranges, or chocolate within 24 hours prior to and after dosing;
21. History of human immunodeficiency virus (HIV) or hepatitis C virus or a positive test at screening for HIV antibody, hepatitis C antibody, or hepatitis B surface antigen;
22. Cumulative blood donation of >500 mL within 2 months prior to the Screening Visit;
23. Use of any prescription or non-prescription medication, including vitamins or herbal medications, within 7 days, or 5 half-lives (if known), whichever is longer, prior to dosing in any of the 3 periods and within 24 hours after dosing in any period. The use of acetaminophen, naproxen, and ibuprofen is permitted except for within 24 hours prior to dosing;
24. Use of any prescription or non-prescription medication that may cause QT prolongation within 14 days, or 5 half lives, whichever is longer, prior to dosing in Period 1 through 24 hours following dosing in Period 3;
25. Any known exposure to prescription or non prescription medications or other substances, such as paint solvents or pesticides, known to induce or inhibit drug metabolizing enzymes or transport system enzymes, within 30 days or 5 half-lives, whichever is longer, prior to dosing in Period 1 through 24 hours following dosing in Period 3, with the exception of hormonal contraception;
26. Unwillingness to abstain from strenuous exercise (e.g., heavy lifting, weight training, calisthenics, aerobics) for at least 48 hours prior to admission to the investigational site;
27. Investigational site personnel directly affiliated with this study;
28. Poor mental function or any other reason to expect subject difficulty in complying with the requirements of the study in the judgment of the Investigator; or
29. Failure to comply with protocol requirements or whose further participation in the study would be unsuitable to the subject, as determined by the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of a therapeutic dose of an IV infusion of eravacycline (TP-434) on cardiac repolarization compared to placebo | 11 weeks
  Calculating the differences between time-matched mean change from baseline of QTcI (ΔΔQTcI = ΔQTcI[TP-434]-ΔQTcI[placebo]) in healthy male and female subjects.

SECONDARY OUTCOMES:
Evaluate the effect of eravacycline (TP-434) on cardiac repolarization | 11 weeks
  * To evaluate the effect of eravacycline (TP-434) on cardiac repolarization compared with placebo by calculating the differences between the time-matched mean changes from baseline of QTcB (ΔΔQTcB) and QTcF (ΔΔQTcF) in healthy male and female subjects;
  * To evaluate the correlation between the differences in time-matched baseline-adjusted mean changes of QTc in eravacycline (TP-434) and placebo (ΔΔQTcI, ΔΔQTcB, and ΔΔQTcF) and plasma concentrations of eravacycline (TP-434), TP-498, and TP-6208;
  * To evaluate the correlation between QTcI, QTcB, and QTcF changes from baseline (ΔQTcI, ΔQTcB, and ΔQTcF) and plasma concentrations of eravacycline (TP-434), TP 498, and TP-6208; and
  * To evaluate assay sensitivity by measuring the effect of moxifloxacin on QTc compared to placebo (ΔΔQTcI).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T Horn, MD, PhD, Study Director — Tetraphase Pharmaceuticals, Inc